CLINICAL TRIAL: NCT04307381
Title: An Open-Label Extension Study of ISIS 721744 in Patients With Hereditary Angioedema
Brief Title: An Extension Study of Donidalorsen (IONIS-PKK-LRx) in Participants With Hereditary Angioedema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 721744-CS3; 2020-000197-14 (EudraCT Number)
Expanded Access: NCT06415448 (Available)
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Hereditary Angioedema
Keywords: Hereditary Angioedema; HAE
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — donidalorsen; IONIS-PKK-LRx

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Donidalorsen (Experimental): Participants will be administered donidalorsen SC for up to 53 weeks. Participants will also be administered donidalorsen in the extended treatment period for an additional 156 weeks, up to week 209.
  Interventions: Drug: Donidalorsen

INTERVENTIONS:
Drug: Donidalorsen — Donidalorsen administered SC
  Other Names: ISIS 721744; IONIS-PKK-LRx

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of extended dosing of donidalorsen administered subcutaneously (SC), with alternative dosing and/or dose frequency with donidalorsen in participants with hereditary angioedema (HAE).

DETAILED DESCRIPTION:
This is an open-label extension study of donidalorsen in up to 24 participants with HAE. The length of participation in the study is approximately 68 weeks, which includes an up to 4-week qualification period, a 52-week treatment period, and a 12-week post-treatment period. Following the Week 53 treatment period visit, participants will receive donidalorsen in an extended treatment period for up to an additional 156 weeks. Participants taking part in the extended treatment period will enter the 12-week post-treatment period after completion of, or early termination from, the extended treatment period.

This study was extended to allow participants to receive donidalorsen for an additional 156 weeks following the initial 53-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Satisfactory completion of ISIS 721744-CS2 (index study) through Week 17 with an acceptable safety and tolerability profile, per Sponsor and Investigator judgement
2. Able and willing to participate in a 64-week study
3. Females must be non-pregnant, non-lactating and either surgically sterile or post-menopausal
4. Males must be surgically sterile or abstinent* or if engaged in sexual relations with a female of child-bearing potential, participant is utilizing an acceptable contraceptive method
5. Participants must have access to, and the ability to use, ≥ 1 acute medication(s) (e.g., plasma-derived or recombinant C1- inhibitor (C1-INH) concentrate or a bradykinin-2 [BK-2] antagonist) to treat angioedema attacks

Exclusion Criteria:

1. Have any new condition or worsening of an existing condition or change or anticipated change in medication, which in the opinion of the Investigator would make the participant unsuitable for enrollment, or could interfere with the participant participating in or completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with at Least One Treatment-emergent Adverse Event (TEAE), Graded by Severity | Up to Week 221

SECONDARY OUTCOMES:
The Time-normalized HAE Attacks (per Month) by Treatment | Up to Week 221
Plasma Prekallikrein (PKK) Levels | Up to Week 221
Consumption of On-demand Medications | Up to Week 221
Angioedema Quality of Life (AE-QoL) Questionnaire Score | Up to Week 221
  The AE-QoL was developed to measure health-related quality of life (HRQoL) impairment in participants with recurrent angioedema. The AE-QoL is a self-administered questionnaire that can be completed in less than 5 minutes. It comprises 17 items across 4 domains: functioning, fatigue/mood, fears/shame, and food. Responses use a 5-point Likert scale ranging from 'never' to 'very often.' Global and domain scores range from 0 to 100, with higher scores indicating greater impairment

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - Ionis Investigative Site, Scottsdale, Arizona
  - Ionis Investigative Site, Santa Monica, California
  - Ionis Investigative Site, Plymouth, Minnesota
  - Ionis Investigative Site, Cincinnati, Ohio
  - Ionis Investigative Site, Hershey, Pennsylvania
  - Ionis Investigative Site, Dallas, Texas
- Ionis Investigative Site, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.
URL: https://vivli.org/ourmember/ionis/

REFERENCES:
- [Derived] Petersen RS, Bordone L, Riedl MA, Tachdjian R, Craig TJ, Lumry WR, Manning ME, Bernstein JA, Raasch J, Zuraw BL, Deng Y, Newman KB, Alexander VJ, Lui C, Schneider E, Cohn DM. A phase 2 open-label extension study of prekallikrein inhibition with donidalorsen for hereditary angioedema. Allergy. 2024 Mar;79(3):724-734. doi: 10.1111/all.15948. Epub 2023 Nov 27. PMID 38009241